CLINICAL TRIAL: NCT03455491
Title: Multicenter Double-blinded Placebo-Controlled Parallel-Group Randomized Clinical Trial of Efficacy, Safety and Choice of an Optimum Dose of XC221 in the Treatment of Influenza and Other Acute Respiratory Viral Infections in Adults
Brief Title: Study to Assess Efficacy and Safety of XC221 in the Treatment of Influenza and Other Acute Respiratory Viral Infections
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PHARMENTERPRISES LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ARI-XC221-02
Record Dates: First submitted 2018-02-28; First posted 2018-03-06 (Actual); Results first posted 2019-11-04 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Acute Respiratory Viral Infections; Influenza
MeSH Terms: conditions — Influenza, Human | interventions — XC221

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Blinding will carried out by using Placebo equivalent to XC221 tablets without active substance and the corresponding labeling of the study drug.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- XC221 100 mg (Experimental): XC221 100 mg orally.
  1 tablet of XC221 100 mg +1 tablet of Placebo 100 mg (in total 2 tablets) once daily during 3 days of treatment period
  Interventions: Drug: XC221 100 mg
- XC221 200 mg (Experimental): XC221 200 mg orally. 2 tablets of XC221 100 mg once daily during 3 days of treatment period
  Interventions: Drug: XC221 200 mg
- Placebo (Placebo Comparator): Placebo orally. 2 tablets of Placebo 100 mg once daily during 3 days of treatment period
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: XC221 100 mg — once daily during 3 days.
  Arms: XC221 100 mg
Drug: XC221 200 mg — once daily during 3 days.
  Arms: XC221 200 mg
Drug: Placebo — once daily during 3 days.
  Arms: Placebo

SUMMARY:
A multicenter double-blinded, randomized, placebo-controlled, parallel-group comparative Phase II clinical study to assess safety, tolerability, efficacy and optimal dose of XC221 vs. placebo in patients with uncomplicated influenza or other ARVI during a 3-day treatment.

The primary objective of the study is to demonstrate the difference in time before the onset of a sustained improvement in clinical symptoms according to the Modified Jackson Scale for ARVI and to determine the optimal dose of XC221 in the treatment of influenza and other ARVI.

DETAILED DESCRIPTION:
11 Russian centers were planned for participation in this study. The study consists of three periods: screening, treatment and follow-up.

All eligible patients will be randomized into 3 groups (groups A, B and C) in a 1:1:1 ratio:

Group A - XC221 100 mg daily (40 patients); Group B - XC221 200 mg daily (40 patients); Group C - Placebo (40 patients).

During the treatment period (3 days), patients will receive XC221 / placebo daily on a background of standard symptomatic therapy. The follow-up period lasts for 11 days.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 18 to 45 years (inclusively).
2. Clinically diagnosed influenza or ARVI.
3. Patient's body temperature ≥37.5ºС and at least 1 symptom from Modified Jackson Scale estimated more than 2 points.
4. Uncomplicated course of influenza or ARVI based on clinical estimations.
5. The first 36 hours from the beginning of symptoms of influenza or ARVI.
6. Women of reproductive age (who are not in menopause and who have not undergone surgical sterilization) and men who have sexual activity should use a reliable method of contraception (acceptable methods of contraception in this study are: intrauterine devices, oral contraceptives, contraceptive patch, long-acting injectable contraceptives, a double barrier method (condom and diaphragm with spermicide) throughout the study period.
7. Compliance with the treatment regimen, visits and laboratory examinations provided by the protocol.
8. Signed Informed Consent Form.

Exclusion Criteria:

1. Existence of complications of influenza or ARVI (including the presence / development of bacterial infection).
2. Hypersensitivity to excipients of the drug XC221 or placebo.
3. Antiviral medications in 7 days prior to screening (antiviral agents, interferons and interferon inducers, drugs that have immunomodulating action) or anti-infective agents of systemic or local action.
4. Severe infection with signs of cardiovascular insufficiency development and other manifestations of infectious-toxic shock, as well as with the presence of neuroinfection syndrome (encephalic and meningoencephalic reactions, polyradiculoneuritis, neuritis).
5. Signs of the development of viral pneumonia (the presence of two or more of the following symptoms): dyspnea, chest pain when coughing, systemic cyanosis, dullness of percussion sound with a symmetrical evaluation of the upper and lower sections of the lungs).
6. Infectious diseases during the last week before including into the study.
7. History of bronchial asthma.
8. History of increased convulsive activity.
9. Severe, decompensated or unstable somatic diseases (any diseases or conditions that are life-threatening or may worsen the patient's prognosis, and make him/her ineligible for the clinical study).
10. History of oncological diseases, HIV, tuberculosis.
11. Diabetes mellitus.
12. Drug or alcohol abuse.
13. Participation in any other clinical trial in the last 90 days.
14. Pregnancy or lactation.
15. Military or prison populations.
16. Impossibility or inability to comply with the study procedures.
17. A member of the investigator's family or other person interested in the results of the study.
18. Abnormal laboratory results, which, according to the study doctor, interfere with the patient's inclusion in the study.
19. History of renal insufficiency.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2018-06-28 (Actual); Study Completion 2018-06-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- Russia (11):
  - City Clinical Hospital №9, Izhevsk
  - Kuban State Medical University, Krasnodar
  - City Clinical Hospital №1 n.a. Semashko, Rostov-on-Don
  - Ryazan State Medical University n.a. Pavlov, Ryazan
  - The Center for Prevention and Fight about AIDS and Infectious Diseases, Saint Petersburg
  - The Consulting and Diagnostic Center with out-patient help of the Administration of the President of the Russian Federation, Saint Petersburg
  - Research Institute of Influenza, Saint Petersburg
  - City Clinical Hospital №40 of Kurortny District, Saint Petersburg
  - Mordovia State Medical University n.a. N.P.Ogarev, Clinical site - Republic Infectious Clinical Hospital, Saransk
  - Volgograd State Medical University, Clinical site - Infectious Regional Clinical Hospital № 1, Volgograd
  - Сlinical Hospital №3, Yaroslavl

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients receiving both in- and outpatient treatment could be enrolled.
Pre-assignment Details: A total of 121 patients were screened to participate in the trial; one patient was withdrawn at screening.
  120 patients were randomly assigned into 3 groups.
Groups:
- Group A: XC221 100 mg orally.
  1 tablet of XC221 100 mg +1 tablet of Placebo 100 mg (in total 2 tablets) once daily during 3 days of treatment period
  XC221 100 mg: once daily during 3 days.
- Group B: XC221 200 mg orally. 2 tablets of XC221 100 mg once daily during 3 days of treatment period
  XC221 200 mg: once daily during 3 days.
- Group C: Placebo orally. 2 tablets of Placebo 100 mg once daily during 3 days of treatment period
  Placebo: once daily during 3 days.
Period: Overall Study
Arm/Group | Group A | Group B | Group C
Started | 40 | 40 | 40
Completed | 40 | 40 | 40
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Group C | Total
Number analyzed (Participants) | 40 | 40 | 40 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 30 (7.3) | 31.1 (7.1) | 32.2 (8.1) | 31.1 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 24 | 23 | 72
  Male | 15 | 16 | 17 | 48
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 40 | 39 | 40 | 119
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Russia | 40 | 40 | 40 | 120
Presence of confirmed viral infection by PCR [Count of Participants; unit: Participants]
  Viral infection confirmed by PCR | 29 | 27 | 22 | 78
  No viral infection confirmed by PCR | 11 | 13 | 18 | 42

OUTCOME MEASURES:

1. Primary Outcome: Time to Sustained Improvement in Clinical Symptoms Based on Modified Jackson Scale for ARVI
Description: The time before the onset of sustained improvement in clinical symptoms according to the Modified Jackson Scale (no more than 1 point for each symptom), measured in hours from the moment of the first dose of the drug.
  Modified Jackson Scale measures individuals' subjective ratings the severity of 12 respiratory symptoms. Ranges for each symptom: 0 points (no symptoms) - 3 points (the most severe). Total score (ranges from 0 to 32 points) is a sum of the point for each symptom.
Time Frame: From the time of randomization up to Day 14
Population: Full Analysis Set (FAS) population
Measure: Median (95% Confidence Interval); unit: hours
Groups:
- XC221 100 mg: XC221 100 mg orally.
  1 tablet of XC221 100 mg +1 tablet of Placebo 100 mg (in total 2 tablets) once daily during 3 days of treatment period
  XC221 100 mg: once daily during 3 days.
Arm/Group | XC221 100 mg | XC221 200 mg | Placebo
Number analyzed (Participants) | 40 | 40 | 40
hours | 57.38 [53.31 to 73.53] | 67.75 [53.69 to 73.87] | 69.64 [63.56 to 88.97]
Statistical Analysis 1: Comparison: XC221 100 mg vs XC221 200 mg vs Placebo; Test type: Superiority; p = 0.3541, Gekhan-Wilcoxon test

2. Secondary Outcome: Time to Body Temperature Normalization
Description: Time to body temperature normalization since treatment initiation, measured in hours (normalization is regarded as setting of body temperature below 37°C without elevation above these values)
Time Frame: From the time of randomization assessed up to Day 14
Population: FAS population
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | XC221 100 mg | XC221 200 mg | Placebo
Number analyzed (Participants) | 40 | 40 | 40
hours | 61.08 (52.85) | 52.26 (34.08) | 61.40 (38.06)
Statistical Analysis 1: Comparison: XC221 100 mg vs XC221 200 mg vs Placebo; Test type: Superiority; p = 0.3597, Gekhan-Wilcoxon test

3. Secondary Outcome: Percentage of Patients With Complications
Description: The percentage of patients with complications of influenza/acute viral URI
Time Frame: From the time of randomization up to Day 14
Population: FAS population
Measure: Count of Participants; unit: Participants
Arm/Group | XC221 100 mg | XC221 200 mg | Placebo
Number analyzed (Participants) | 40 | 40 | 40
Participants
  No complications | 39 | 40 | 40
  With complications | 1 | 0 | 0

4. Secondary Outcome: The Area Under the Curve "Modified Jackson Scale Score" During 3-day Therapy
Description: Modified Jackson Scale measures individuals' subjective ratings the severity of 12 respiratory symptoms. Ranges for each symptom: 0 points (no symptoms) - 3 points (the most severe). Total score (ranges from 0 to 32 points) is a sum of the point for each symptom.
Time Frame: From randomization up to 3 days of treatment
Population: FAS population
Measure: Mean (Standard Deviation); unit: Ln(units_on_a_scale*sec)
Arm/Group | XC221 100 mg | XC221 200 mg | Placebo
Number analyzed (Participants) | 40 | 40 | 40
Ln(units_on_a_scale*sec) | 14.6 (0.4) | 14.6 (0.4) | 14.7 (0.4)
Statistical Analysis 1: Comparison: XC221 100 mg vs XC221 200 mg vs Placebo; Test type: Superiority; p = 0.4551, ANOVA; one-way ANOVA

ADVERSE EVENTS:
Time Frame: 16 days
Arm/Group | Group A | Group B | Group C
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 16/40 | 13/40 | 14/40
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=40) | Group B (N=40) | Group C (N=40)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Strengthening cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Epigastric pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Loose stools (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Bacterial tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Labial herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Basophilia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 1 (1)
Hoarseness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Tickling (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhea (Ear and labyrinth disorders) | 1 (1) | 2 (2) | 1 (1)
Increased nasal congestion (Ear and labyrinth disorders) | 2 (2) | 2 (2) | 3 (3)
Increased hoarseness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Tickering (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (2)
Strengthening rhinorrhea (Ear and labyrinth disorders) | 3 (3) | 2 (2) | 5 (5)
Increased sneezing (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 1 (1)
Sneezing (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 2 (2) | 4 (4)
Strengthening headache (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Strengthening myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Tearing (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Hypothermia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fever (General disorders) | 3 (4) | 2 (2) | 2 (3)
Chill increase (General disorders) | 1 (1) | 1 (1) | 1 (1)
Malaise (General disorders) | 1 (1) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0)
Periodic temperature rise (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fever increase (General disorders) | 4 (4) | 3 (3) | 2 (3)
Strengthening ailments (General disorders) | 5 (5) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-25): https://cdn.clinicaltrials.gov/large-docs/91/NCT03455491/Prot_SAP_000.pdf